CLINICAL TRIAL: NCT00268996
Title: An International, Multicenter, Randomized, Placebo-controlled, Parallel-group, 1 Year Treatment, Integrated Biomarkers and Imaging Study in Subjects With Angiographically Documented Coronary Heart Disease (CHD) to Examine the Effects of the Novel Lipoprotein-associated Phospholipase A2 (Lp-PLA2) Inhibitor SB-480848 on Intermediate Cardiovascular Endpoints, Patient Safety and Tolerability
Brief Title: Integrated Biomarker And Imaging Study - 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB-480848/026
Record Dates: First submitted 2005-12-21; First posted 2005-12-23 (Estimated); Results first posted 2018-02-19 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2017-08

CONDITIONS: Atherosclerosis
Keywords: Coronary artery disease; Lipoprotein-associated Phospholipase A2; palpography; hs-CRP; endothelial function; intravascular ultrasound
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease | interventions — darapladib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Subjects with ACS and evidence of MN:SB-480848 (Experimental): Enrolled subjects (subjects with ACS and evidence of myocardial necrosis) will receive 160mg of SB-480848 once daily with food for 52 weeks
  Interventions: Drug: SB-480848
- Subjects with ACS and evidence of MN: placebo (Placebo Comparator): Enrolled subjects (subjects with ACS and evidence of myocardial necrosis) will receive SB-480848 matching placebo once daily with food for 52 weeks
  Interventions: Drug: SB-480848 matching placebo
- Non-ACS and ACS subjects without evidence of MN: SB-480848 (Experimental): Enrolled subjects (non-ACS subjects and those ACS subjects without evidence of myocardial necrosis) will receive 160mg of SB-480848 once daily with food for 52 weeks
  Interventions: Drug: SB-480848
- Non-ACS and those ACS subjects without evidence of MN: placebo (Placebo Comparator): Enrolled subjects (non-ACS subjects and those ACS subjects without evidence of myocardial necrosis) will receive SB-480848 matching placebo once daily with food for 52 weeks
  Interventions: Drug: SB-480848 matching placebo

INTERVENTIONS:
Drug: SB-480848 — SB-480848 is available as enteric-coated, free-base micronized tablet
  Arms: Non-ACS and ACS subjects without evidence of MN: SB-480848; Subjects with ACS and evidence of MN:SB-480848
Drug: SB-480848 matching placebo — Placebo is available as enteric-coated, free-base micronized tablet
  Arms: Non-ACS and those ACS subjects without evidence of MN: placebo; Subjects with ACS and evidence of MN: placebo

SUMMARY:
IBIS-2 is a study using SB-480848 versus placebo in subjects with angiographically documented coronary heart disease. Endpoints include coronary imaging, endothelial function, biomarkers, safety and tolerability.

DETAILED DESCRIPTION:
Integrated Biomarker and Imaging Study -2 (IBIS-2): An International, Multicenter, Randomized, Placebo-controlled, Parallel-group, 1 Year Treatment, Integrated Biomarkers and Imaging Study in Subjects with Angiographically Documented Coronary Heart Disease (CHD) to Examine the Effects of the Novel Lipoprotein-associated Phospholipase A2 (Lp-PLA2) inhibitor SB-480848 on Intermediate Cardiovascular Endpoints, Patient Safety and Tolerability.

ELIGIBILITY:
Inclusion criteria:

* Successful PCI (Percutaneous Coronary Intervention) or uncomplicated diagnostic catheterization
* Suitable non-intervened coronary artery with IVUS
* Antiplatelet therapy

Exclusion criteria:

* Clinical instability
* Previous CABG (Coronary Artery By-pass Graft) surgery
* Planned major surgery
* Recent stroke
* Abnormal QTc
* Renal or hepatic impairment
* Uncontrolled hypertension
* Use of corticosteroids
* Class III or IV heart failure
* Asthma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2005-11-10 (Actual); Primary Completion 2007-08-28 (Actual); Study Completion 2007-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- GSK Investigational Site, Vienna, Austria
- Belgium (3):
  - GSK Investigational Site, Aalst
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Liège
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, Aarhus N, Denmark
- France (2):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Brest
- Germany (7):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Ulm, Baden-Wurttemberg
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bad Nauheim, Hesse
  - GSK Investigational Site, Essen, North Rhine-Westphalia
  - GSK Investigational Site, Bad Segeberg, Schleswig-Holstein
  - GSK Investigational Site, Hamburg
- Netherlands (4):
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Leeuwarden
  - GSK Investigational Site, Rotterdam
- GSK Investigational Site, Bergen, Norway
- Poland (2):
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
- Spain (2):
  - GSK Investigational Site, Marid
  - GSK Investigational Site, Santander
- GSK Investigational Site, Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Serruys PW, Garcia-Garcia HM, Buszman P, Erne P, Verheye S, Aschermann M, Duckers H, Bleie O, Dudek D, Botker HE, von Birgelen C, D'Amico D, Hutchinson T, Zambanini A, Mastik F, van Es GA, van der Steen AF, Vince DG, Ganz P, Hamm CW, Wijns W, Zalewski A; Integrated Biomarker and Imaging Study-2 Investigators. Effects of the direct lipoprotein-associated phospholipase A(2) inhibitor darapladib on human coronary atherosclerotic plaque. Circulation. 2008 Sep 9;118(11):1172-82. doi: 10.1161/CIRCULATIONAHA.108.771899. Epub 2008 Sep 1. PMID 18765397
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: SB-480848/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: SB-480848/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: SB-480848/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: SB-480848/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: SB-480848/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: SB-480848/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: SB-480848/026 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in participants with angiographically documented coronary artery disease (CHD) at 23 sites in 10 countries. The study was initiated on 10 November 2005 and completed on 28 August 2007.
Pre-assignment Details: There were 451 participants screened for enrollment of whom 121 failed screening. A total of 330 participants were randomized to receive treatment. Among the randomized participants, 4 from placebo arm and 3 from darapladib arm did not receive study drug. The remaining 323 participants received at least one dose of study drug.
Groups:
- Placebo: Eligible participants received the matching placebo for 52 weeks. Participants were instructed to administer one tablet (swallowed intact and not chewed) in the morning each day with food.
- Darapladib 160mg EC Tablet: Eligible participants received SB-480848 (darapladib) 160 milligram (mg) enteric coated (EC) tablets once daily for 52 weeks. Participants were instructed to administer one tablet (swallowed intact and not chewed) in the morning each day with food.
Period: Overall Study
Arm/Group | Placebo | Darapladib 160mg EC Tablet
Started | 151 | 172
Completed | 130 | 152
Not Completed | 21 | 20
Not completed — Adverse Event | 11 | 7
Not completed — Lost to Follow-up | 3 | 1
Not completed — Withdrawal by Subject | 5 | 11
Not completed — Non-compliance | 1 | 0
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Darapladib 160 mg EC Tablet: Eligible participants received darapladib 160 mg EC tablet once daily for 52 weeks. Participants were instructed to administer one tablet (swallowed intact and not chewed) in the morning each day with food.
- Total: Total of all reporting groups
Arm/Group | Placebo | Darapladib 160 mg EC Tablet | Total
Number analyzed (Participants) | 151 | 172 | 323
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.3 (10.86) | 59.4 (9.81) | 58.4 (10.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 32 | 57
  Male | 126 | 140 | 266
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 146 | 171 | 317
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Circulating High Sensitivity C- Reactive Protein (Hs-CRP) Levels at Week 52.
Description: hs-CRP is a pentameric protein that is rapidly upregulated in response to inflammation and tissue damage and assessed as circulating biomarkers associated with atherosclerosis and cardiovascular risk. Last Observation Carried Forward (LOCF) data was reported. Only data from 3 months onwards was carried forward. hs-CRP has a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of hs-CRP levels at Week 52 were reported. The levels were analyzed using analysis of co-variance (ANCOVA), with Acute Coronary Syndrome (ACS) status, pooled country and treatment included as covariates.
Time Frame: Week 52
Population: The biomarker evaluable population was comprised of all randomized participants who received at least one dose of study drug, with an evaluable biomarker assessment at 3 months (Day 77) or later.
Measure: Geometric Mean (95% Confidence Interval); unit: mg per litre (mg/L)
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 140 | 162
mg per litre (mg/L) | 1.034 [0.854 to 1.251] | 0.913 [0.765 to 1.090]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.348, ANCOVA; Adjusted percentage change = -11.717, 95% CI 2-sided [-31.995 to 14.607] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet /Placebo) - 1 multiplied by 100]

2. Primary Outcome: Change From Baseline in the Density of Rotterdam Classification (ROC) Grade III/IV Strain Spots/10 Millimeter (mm) Within the Region of Interest (ROI) on IVUS Grey Scale Based Palpography at the End of Week 52.
Description: The ROC grade III/IV strain spots per 10 millimetre (mm) within the ROI on intravascular ultrasound (IVUS) grey scale based palpography were assessed and change from Baseline at end of 52 was reported. Change from Baseline was calculated as the density of spots at the end of study minus the density of spots recorded at Baseline. If either value was considered missing then the change from Baseline value was missing for the participant. Between treatment group comparisons of change from Baseline were analyzed using ANCOVA adjusting for ACS status, pooled country, Baseline value, matched segment length and treatment. Adjusted means and associated standard errors for each treatment group were presented. The baseline value for each participant was defined as the last value prior to the first dose of study drug.
Time Frame: Baseline and Week 52
Population: The imaging evaluable population was comprised of all randomized participants who received at least one dose of study drug, with an evaluable baseline and end of treatment imaging assessment at 6 months (Day 154) or later. The participants available at the time of assessment were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: Spots/10 mm
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 115 | 131
Spots/10 mm | 0.003 (0.048) | -0.079 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.220, ANCOVA; Adjusted Treatment Difference = -0.082, 95% CI 2-sided [-0.214 to 0.049] — Difference in adjusted means is shown (Darapladib 160 mg EC tablet - Placebo)

3. Secondary Outcome: Circulating Hs-CRP at the End of Week 26.
Description: hs-CRP is a pentameric protein that is rapidly upregulated in response to inflammation and tissue damage and assessed as circulating biomarkers associated with atherosclerosis and cardiovascular risk. LOCF data was reported. Only data from 3 months onwards was carried forward. hs-CRP has a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of hs-CRP levels at Week 26 were reported. The levels were analyzed using ANCOVA, with ACS status, pooled country and treatment included as covariates.
Time Frame: Week 26
Population: Biomarker evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 140 | 162
mg/L | 0.924 [0.774 to 1.102] | 0.960 [0.815 to 1.131]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.751, ANCOVA; Adjusted percentage change = 3.977, 95% CI 2-sided [-18.331 to 32.379] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet /Placebo) - 1 multiplied by 100]

4. Secondary Outcome: Mean Lipoprotein Phospholipase A2 (Lp-PLA2) Activity at the End of Week 26 and Week 52
Description: Lp-PLA2 is a calcium-independent phospholipase A2 enzyme associated with low density lipoprotein (LDL) in plasma. Blood samples were collected at baseline and at Week 4, 13, 26, and 52 and Lp-PLA2 activity was determined. Percentage inhibition of Lp-PLA2 activity relative to baseline was calculated as, percent inhibition = ([baseline value - post baseline value] x 100) / baseline value. The baseline value for each participant was defined as the last value prior to the first dose of study drug.
Time Frame: Week 26 and Week 52
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: micromole per minute per Litre
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 140 | 162
micromole per minute per Litre
  Week 26 LOCF | 151.412 [143.592 to 159.657] | 59.449 [56.591 to 62.452]
  Week 52 LOCF | 152.061 [144.109 to 160.452] | 61.850 [58.838 to 65.015]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet at Week 26 (LOCF); Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted percentage change = -60.737, 95% CI 2-sided [-63.486 to -57.780] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet /Placebo) - 1 multiplied by 100]
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet at Week 52 (LOCF); Test type: Superiority or Other; p < 0.001, ANCOVA; Adjusted percentage change = -59.326, 95% CI 2-sided [-62.210 to -56.222] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet /Placebo) - 1 multiplied by 100]

5. Secondary Outcome: Change From Baseline in Plaque Volume as IVUS-Grey Scale Assessments at Week 52
Description: Change from Baseline was calculated for each IVUS grey scale assessment recorded at the end of study. The Baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from Baseline was calculated as plaque volume at Week 52 minus Baseline value. The data was analyzed using ANCOVA, with ACS status, pooled country, Baseline value, matched segment length and treatment included as covariates.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population
Measure: Least Squares Mean (Standard Error); unit: Cubic millimetre (mm^3)
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 118 | 143
Cubic millimetre (mm^3) | -5.126 (2.715) | -4.873 (2.464)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.945, ANCOVA; Adjusted Treatment Difference = 0.253, 95% CI 2-sided [-6.998 to 7.504] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet - Placebo)

6. Secondary Outcome: Change From Baseline in Percent Obstruction Volume as IVUS-Grey Scale Assessments at Week 52
Description: Change from Baseline in percent obstruction volume was calculated for each IVUS grey scale assessment recorded. Percent obstruction volume was calculated as (Plaque volume/ Vessel volume *100). The Baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from Baseline was calculated as plaque volume at Week 52 minus Baseline value. The data was analyzed using ANCOVA, with ACS status, pooled country, baseline value, matched segment length and treatment included as covariates.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population
Measure: Least Squares Mean (Standard Error); unit: Percentage of mm^3
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 118 | 143
Percentage of mm^3 | 0.007 (0.354) | -0.054 (0.321)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.898, ANCOVA; Difference in adjusted means = -0.062, 95% CI 2-sided [-1.009 to 0.886] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet - Placebo)

7. Secondary Outcome: Change From Baseline in Necrotic Core Volume as Intravenous Ultrasound-Virtual Histology (IVUS-VH) Assessments at Week 52
Description: Change from Baseline was calculated for each IVUS-VH assessment recorded at the end of study. The necrotic core volume was calculated as mean necrotic area multiplied by mean of Baseline and follow-up length. Change from Baseline was calculated as plaque volume at Week 52 minus Baseline value. The data was analyzed using ANCOVA, with ACS status, pooled country, Baseline value, matched segment length and treatment included as covariates. The Baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from Baseline in necrotic core volume as IVUS-VH assessments at Week 52 was reported.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 110 | 129
mm^3 | 4.633 (1.491) | -0.531 (1.376)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.012, ANCOVA; Difference in adjusted means = -5.165, 95% CI 2-sided [-9.185 to -1.145] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet - Placebo)

8. Secondary Outcome: Change From Baseline in Necrotic Core as a Percent of IVUS-VH Plaque at the End of Week 52.
Description: Change from baseline was calculated for each IVUS-VH assessment recorded at the end of study. The baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from baseline in percent necrotic core was calculated as percent necrotic core at Week 52 minus baseline value. The data was analyzed using ANCOVA, with ACS status, pooled country, baseline value, matched segment length and treatment included as covariates. Change from Baseline in necrotic core as a percent of IVUS-VH plaque at the end of week 52 was reported.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population
Measure: Least Squares Mean (Standard Error); unit: Percent Necrotic core
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 110 | 129
Percent Necrotic core | 2.502 (0.722) | 0.535 (0.666)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.047, ANCOVA; Difference in adjusted means = -1.967, 95% CI 2-sided [-3.912 to -0.022] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet - Placebo)

9. Secondary Outcome: Mean Interlukin 6 (IL-6) Levels as Circulating Biomarkers Associated With Inflammatory Burden at Week 26 and Week 52
Description: Blood was collected at baseline, Week 4, 13, 26 and 52 for evaluation of biomarkers. Mean IL-6 levels as circulating biomarkers associated with inflammatory burden at Week 26 and Week 52 were assessed and reported. LOCF data was reported. Only data from 3 months onwards was carried forward. IL-6 had a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of IL-6 levels at Week 26 and 52 were reported. The levels were analyzed using ANCOVA, with ACS status, pooled country and treatment included as covariates.
Time Frame: Week 26 and Week 52
Population: Biomarker evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per litre (ng/L)
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 140 | 162
Nanograms per litre (ng/L)
  Week 26 LOCF: number analyzed (Participants) | 135 | 160
  Week 26 LOCF | 1.851 [1.609 to 2.128] | 1.979 [1.741 to 2.250]
  Week 52 LOCF: number analyzed (Participants) | 137 | 161
  Week 52 LOCF | 2.019 [1.749 to 2.331] | 2.267 [1.985 to 2.588]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Week 26 (LOCF): Comparison between Placebo vs Darapladib 160 mg EC tablet; Test type: Superiority or Other; p = 0.487, ANCOVA; Adjusted percentage change = 6.958, 95% CI 2-sided [-11.568 to 29.364] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet /Placebo) - 1 multiplied by 100]
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Week 52 (LOCF): Comparison between Placebo Vs Darapladib 160 mg EC tablet; Test type: Superiority or Other; p = 0.247, ANCOVA; Adjusted percentage change = 12.255, 95% CI 2-sided [-7.725 to 36.562] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet /Placebo) - 1 multiplied by 100]

10. Secondary Outcome: Mean Intercellular Adhesion Molecule-1 (ICAM-1) Levels as Circulating Biomarkers Associated With Inflammatory Burden at Week 26 and Week 52
Description: Blood was collected at baseline, Week 4, 13, 26 and 52 for evaluation of biomarkers. Mean ICAM-1 levels as circulating biomarkers associated with inflammatory burden at Week 26 and Week 52 were assessed and reported. LOCF data was reported. Only data from 3 months onwards was carried forward. ICAM-1 had a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of ICAM-1 levels at Week 26 and 52 were reported. The levels were analyzed using ANCOVA, with ACS status, pooled country and treatment included as covariates.
Time Frame: Week 26 and Week 52
Population: Biomarker evaluable population.
Measure: Geometric Mean (95% Confidence Interval); unit: nanogram per millilitre (ng/mL)
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 140 | 161
nanogram per millilitre (ng/mL)
  Week 26 (LOCF) | 269.444 [258.932 to 280.383] | 266.447 [256.744 to 276.516]
  Week 52 (LOCF) | 277.947 [265.822 to 290.624] | 268.950 [257.998 to 280.367]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 26 (LOCF); Test type: Superiority or Other; p = 0.687, ANCOVA; Adjusted percentage change = -1.112, 95% CI 2-sided [-6.363 to 4.433] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Test type: Superiority or Other; p = 0.290, ANOVA; Adjusted percentage change = -3.237, 95% CI 2-sided [-8.976 to 2.865] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]

11. Secondary Outcome: Mean Myeloperoxidase (MPO) Levels as Circulating Biomarkers Associated With Inflammatory Burden at Week 26 and Week 52
Description: Blood was collected at baseline, Week 4, 13, 26 and 52 for evaluation of biomarkers. Mean MPO levels as circulating biomarkers associated with inflammatory burden at Week 26 and Week 52 were assessed and reported. LOCF data was reported. Only data from 3 months onwards was carried forward. MPO had a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of MPO levels at Week 26 and 52 were reported. The levels were analyzed using ANCOVA, with ACS status, pooled country and treatment included as covariates.
Time Frame: Week 26 and Week 52
Population: Biomarker evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: picomole per litre (pmol/L)
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 139 | 162
picomole per litre (pmol/L)
  Week 26 (LOCF) | 324.534 [294.535 to 357.589] | 378.811 [346.275 to 414.405]
  Week 52 (LOCF) | 370.999 [331.989 to 414.592] | 405.339 [365.718 to 449.253]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 26 (LOCF); Test type: Superiority or Other; p = 0.022, ANCOVA; Adjusted percentage change = 16.725, 95% CI 2-sided [2.232 to 33.271] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 52 (LOCF); Test type: Superiority or Other; p = 0.252, ANCOVA; Adjusted percentage change = 9.256, 95% CI 2-sided [-6.136 to 27.172] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]

12. Secondary Outcome: Mean sCD40L Levels as Circulating Biomarkers Associated With Inflammatory Burden at Week 26 and Week 52
Description: Blood was collected at baseline, Week 4, 13, 26 and 52 for evaluation of biomarkers. Mean sCD40L levels as circulating biomarker associated with inflammatory burden at Week 26 and Week 52 were assessed and reported. sCD40L had a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of sCD40L levels at Week 26 and 52 were reported. The levels were analyzed using ANCOVA, with ACS status, pooled country and treatment included as covariates.
Time Frame: Week 26 and Week 52
Population: Safety Population comprised of all randomized participants who received at least one dose of study drug. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: pg/ml
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 151 | 172
pg/ml
  Week 26: number analyzed (Participants) | 123 | 132
  Week 26 | 178.738 [152.832 to 209.035] | 206.351 [177.412 to 240.012]
  Week 52: number analyzed (Participants) | 107 | 113
  Week 52 | 183.449 [149.887 to 224.526] | 254.200 [208.840 to 309.412]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 26; Test type: Superiority or Other; p = 0.196, ANCOVA; Adjusted percentage change = 15.449, 95% CI 2-sided [-7.204 to 43.632] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 52; Test type: Superiority or Other; p = 0.024, ANCOVA; Adjusted percentage change = 38.567, 95% CI 2-sided [4.355 to 83.997] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]

13. Secondary Outcome: Mean Matrix Metaloproteinases-9 (MMP-9) Levels as Circulating Biomarkers Associated With Plaque Instability at Week 26 and Week 52.
Description: Blood was collected at baseline, Week 4, 13, 26 and 52 for evaluation of biomarkers. Mean MMP-9 levels as circulating biomarkers associated with plaque instability at Week 26 and Week 52 were assessed and reported. LOCF data was reported. Only data from 3 months onwards was carried forward MMP-9 had a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of MMP-9 levels at Week 26 and 52 were reported. The levels were analyzed using ANCOVA, with ACS status, pooled country and treatment included as covariates.
Time Frame: Week 26 and Week 52
Population: Biomarker evaluable population
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per litre (mcg/L)
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 140 | 162
microgram per litre (mcg/L)
  Week 26 LOCF | 481.581 [429.483 to 539.997] | 471.477 [423.894 to 524.401]
  Week 52 LOCF | 488.998 [432.454 to 552.935] | 498.709 [444.895 to 559.032]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 26 (LOCF); Test type: Superiority or Other; p = 0.790, ANCOVA; Adjusted percentage change = -2.098, 95% CI 2-sided [-16.303 to 14.517] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 52 (LOCF); Test type: Superiority or Other; p = 0.818, ANCOVA; Adjusted percentage change = 1.986, 95% CI 2-sided [-13.807 to 20.673] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]

14. Secondary Outcome: Mean Levels of Oxidised Phospholipids/ Apolipoprotein B100 (oxPL/apoB) Ratio as Target Circulating Biomarkers at the End of Week 26 and Week 52.
Description: Blood was collected at baseline, Week 4, 13, 26 and 52 for evaluation of biomarkers. Mean OXPL/LAPO B levels as circulating biomarkers associated with Lp-PLA2 target-related biomarkers at Week 26 and Week 52 were assessed and reported. LOCF data was reported. Only data from 3 months onwards was carried forward. OXPL/LAPO B had a skewed distribution and values were log transformed before analysis. The statistics was calculated on the log transformed data and back transformed. The adjusted geometric means of OXPL/LAPO B levels at Week 26 and 52 were reported. The levels were analyzed using ANCOVA, with ACS status, pooled country and treatment included as covariates.
Time Frame: Week 26 and Week 52
Population: Biomarker evaluable population.
Measure: Geometric Mean (95% Confidence Interval); unit: Relative light units (RLU)
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 140 | 162
Relative light units (RLU)
  Week 26 LOCF | 3114.718 [2695.797 to 3598.739] | 3106.872 [2716.642 to 3553.156]
  Week 52 LOCF | 2711.118 [2017.411 to 3643.363] | 2478.376 [1883.212 to 3261.634]
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 26 (LOCF); Test type: Superiority or Other; p = 0.980, ANCOVA; Adjusted percentage change = -0.252, 95% CI 2-sided [-18.151 to 21.561] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet once daily at Week 52 (LOCF); Test type: Superiority or Other; p = 0.663, ANCOVA; Adjusted percentage change = -8.585, 95% CI 2-sided [-39.007 to 37.012] — Adjusted percentage change is shown [(Darapladib 160 mg EC tablet once daily/Placebo) - 1 multiplied by 100]

15. Secondary Outcome: Mean Levels of Oxidized Non-esterified Fatty Acids (Ox-NEFA) as Target Circulating Biomarkers at the End of Week 26 and Week 52
Description: Mean ox-NEFA levels as circulating biomarkers associated with Lp-PLA2 target-related biomarkers at Week 26 and Week 52 was planned to be assessed. However, the parameter data were not collected for this endpoint.
Time Frame: Week 26 and Week 52
Population: Biomarker evaluable population
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Change From Baseline in Vessel Volume and Lumen Volume as IVUS-Grey Scale Assessments at Week 52.
Description: Change from baseline in vessel volume and lumen volume calculated for each IVUS grey scale assessment recorded. Vessel volume (i.e., coronary remodelling) defined by the leading edge of echogenic adventitia/external elastic membrane (EEM) and calculated as, mean vessel area multiplied mean of vessel length at Baseline and Follow-up. Lumen volume was circumscribed by the leading edge of intima/plaque and calculated as mean lumen area multiplied by mean lumen length at Baseline and Follow-up. The baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from baseline was calculated as vessel volume or lumen volume at Week 52 minus baseline value.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 118 | 143
mm^3
  Vessel volume | -11.211 (5.400) | -9.453 (4.901)
  Lumen volume | -6.693 (5.160) | -4.066 (4.682)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; For vessel volume; Test type: Superiority or Other; p = 0.811, ANCOVA; Adjusted treatment Difference = 1.758, 95% CI 2-sided [-12.675 to 16.192] — Difference in adjusted means are shown (Darapladib 160mg EC tablet once daily - Placebo)
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; For lumen volume; Test type: Superiority or Other; p = 0.708, ANCOVA; Adjusted Treatment Difference = 2.627, 95% CI 2-sided [-11.171 to 16.425] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet once daily - Placebo)

17. Secondary Outcome: Change From Baseline in Mean Plaque Area, Mean Vessel Area, and Mean Lumen Area as IVUS-Grey Scale Assessments at Week 52.
Description: Change from baseline in was mean plaque area, mean vessel area, and mean lumen area were derived from IVUS system at each IVUS grey scale assessment recorded. The baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from baseline was calculated as mean area of the parameter (plaque/vessel/lumen) at Week 52 minus baseline value. The data was reported based on observed cases. Data analyzed using ANCOVA, with ACS status, pooled country, baseline value, matched segment length and treatment included as covariates.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population
Measure: Least Squares Mean (Standard Error); unit: mm2
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 118 | 143
mm2
  Mean plaque area | -0.112 (0.056) | -0.124 (0.050)
  Mean vessel area | -0.242 (0.115) | -0.194 (0.104)
  Mean lumen area | -0.130 (0.112) | -0.069 (0.101)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet: Mean vessel area; Test type: Superiority or Other; p = 0.873, ANCOVA — Data analyzed using ANCOVA, with ACS status, pooled country, baseline value , matched segment length and treatment included as covariates; Adjusted Treatment Difference = -0.012, 95% CI 2-sided [-0.160 to 0.136] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet one daily - Placebo)
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet: Mean vessel area; Test type: Superiority or Other; p = 0.756, ANCOVA; Data analyzed using ANCOVA, with ACS status, pooled country, baseline value , matched segment length and treatment included as covariates; Adjusted Treatment Difference = 0.048, 95% CI 2-sided [-0.258 to 0.354] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet one daily - Placebo)
Statistical Analysis 3: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet: Mean lumen area; Test type: Superiority or Other; p = 0.687, ANCOVA; [statistical method as in outcome 17, analysis 2]; Adjusted Treatment Difference = 0.061, 95% CI 2-sided [-0.237 to 0.360] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet one daily - Placebo)

18. Secondary Outcome: Change From Baseline in Fibrous Tissue Volume and Fibro-fatty Volume as IVUS-VH Assessments at Week 52
Description: Change from baseline in fibrous tissue volume and fibro-fatty volume were derived from IVUS system at each IVUS grey scale assessment recorded. Fibrous tissue volume was calculated as mean fibro-fatty area multiplied by mean of Baseline and Follow-up length. Fibro-fatty volume was calculated as mean fibrous area multiplied by mean of Baseline and Follow-up length.
  The baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from baseline was calculated as mean Fibrous tissue volume or Fibro-fatty volume at Week 52 minus baseline value. The data was reported based on observed cases. Data analyzed using ANCOVA, with ACS status, pooled country, baseline value , matched segment length and treatment included as covariates.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population
Measure: Least Squares Mean (Standard Error); unit: mm^3
Groups:
- Darapladib 160 mg EC Tablet: Eligible participants received darapladib 160 mg EC tablet one daily for 52 weeks. Participants were instructed to administer one tablet (swallowed intact and not chewed) in the morning each day with food.
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 110 | 129
mm^3
  Fibrous tissue volume | -6.985 (2.312) | -7.569 (2.133)
  Fibro-fatty volume | -3.342 (1.734) | -1.415 (1.600)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet: Fibrous tissue volume; Test type: Superiority or Other; p = 0.854, ANCOVA; Data analyzed using ANCOVA, with ACS status, pooled country, baseline value, matched segment length and treatment included as covariates; Adjusted Treatment Difference = -0.584, 95% CI 2-sided [-6.819 to 5.650] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet one daily - Placebo)
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet: Fibro-fatty volume; Test type: Superiority or Other; p = 0.418, ANCOVA — Data analyzed using ANCOVA, with ACS status, pooled country, baseline value, matched segment length and treatment included as covariates; Adjusted Treatment Difference = 1.926, 95% CI 2-sided [-2.748 to 6.600] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet one daily - Placebo)

19. Secondary Outcome: Change From Baseline in Fibrous Tissue and Fibro-fatty as a Percent of IVUS-VH Plaque as IVUS-VH Assessments at Week 52
Description: Fibro-fatty as percentage of VH plaque and Fibrous tissue as percentage of VH plaque were derived from IVUS-VH system. The baseline value for each participant was defined as the last value prior to the first dose of study drug. Change from baseline was calculated as Fibro-fatty as percentage of VH plaque or Fibrous tissue as percentage of VH plaque at Week 52 minus baseline value. The data was reported based on observed cases. Data analyzed using ANCOVA, with ACS status, pooled country, baseline value , matched segment length and treatment included as covariates.
Time Frame: Baseline and Week 52
Population: Imaging evaluable population
Measure: Least Squares Mean (Standard Error); unit: Percentage of VH
Groups:
- Darapladib 160 mg EC Tablet: Eligible participants received darapladib 160 mg EC tablet for 52 weeks. Participants were instructed to administer one tablet (swallowed intact and not chewed) in the morning each day with food.
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
Number analyzed (Participants) | 110 | 129
Percentage of VH
  Fibrous tissue as percentage of VH plaque | -4.007 (0.631) | -2.007 (0.582)
  Fibro-fatty as percentage of VH plaque | -0.782 (0.881) | -0.043 (0.813)
Statistical Analysis 1: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet: Fibrous tissue as % of VH plaque; Test type: Superiority or Other; p = 0.021, ANOVA; [statistical method as in outcome 18, analysis 1]; Adjusted Treatment Difference = 2, 95% CI 2-sided [0.299 to 3.701] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet one daily - Placebo)
Statistical Analysis 2: Comparison: Placebo vs Darapladib 160 mg EC Tablet; Placebo vs Darapladib 160 mg EC tablet: Fibro-fatty as percentage of VH plaque; Test type: Superiority or Other; p = 0.540, ANCOVA; [statistical method as in outcome 18, analysis 1]; Adjusted Treatment Difference = 0.739, 95% CI 2-sided [-1.635 to 3.114] — Difference in adjusted means are shown (Darapladib 160 mg EC tablet one daily - Placebo)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time a participant consents to participate until completion of follow-up period (10 to 21 days after discontinuation of treatment). On-treatment (up to 52 weeks) serious-AE (SAE) and non-SAE are reported.
Description: Safety population was used for collection of AEs.
Arm/Group | Placebo | Darapladib 160 mg EC Tablet
All-Cause Mortality (participants affected / at risk) | 0/151 | 0/172
Serious Adverse Events (participants affected / at risk) | 45/151 | 46/172
Other Adverse Events (participants affected / at risk) | 37/151 | 59/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=151) | Darapladib 160 mg EC Tablet (N=172)
Angina pectoris (Cardiac disorders) | 9 | 9
Coronary artery disease (Cardiac disorders) | 3 | 12
Acute myocardial infarction (Cardiac disorders) | 4 | 3
Angina unstable (Cardiac disorders) | 4 | 3
In-stent coronary artery restenosis (Cardiac disorders) | 7 | 0
Coronary artery restenosis (Cardiac disorders) | 3 | 1
Coronary artery stenosis (Cardiac disorders) | 2 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0
Arteriospasm coronary (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac asthma (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac pseudoaneurysm (Cardiac disorders) | 1 | 0
Coronary artery dissection (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 2 | 3 — General disorders and administration site conditions
Chest pain (General disorders) | 1 | 0 — General disorders and administration site conditions
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Global amnesia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Cardiac procedure complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 2
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Occult blood positive (Investigations) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Bladder tamponade (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=151) | Darapladib 160 mg EC Tablet (N=172)
Angina pectoris (Cardiac disorders) | 12 (14) | 18 (23)
Urine odour abnormal (Renal and urinary disorders) | 4 (4) | 17 (17)
Abnormal faeces (Gastrointestinal disorders) | 2 (2) | 18 (18)
Fatigue (General disorders) | 10 (11) | 10 (10)
Nasopharyngitis (Infections and infestations) | 10 (12) | 7 (8)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 13 (15)
Non-cardiac chest pain (General disorders) | 7 (7) | 9 (11)
Oedema peripheral (General disorders) | 2 (2) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.